CLINICAL TRIAL: NCT03995823
Title: MRI Evaluation of Nidus Occlusion After Gamma Knife Radiosurgery of Cerebral Arteriovenous Malformations - A Prospective Preliminary Study
Brief Title: Evaluation of Nidus Occlusion After Gamma Knife Radiosurgery of Cerebral Arteriovenous Malformations Using Magnetic Resonance Imaging
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Collaborators: Medical Scientific Fund of the Mayor of Vienna (Other)
Responsible Party: Principal Investigator, Josa M Frischer, MD, PhD, Assoc.Prof.Priv.Doz.Dr.PhD, Medical University of Vienna
Other Study IDs: 1497/2018; 18096 (Other Grant/Funding Number: Medical Scientific Fund of the Mayor of Vienna)
Record Dates: First submitted 2019-06-17; First posted 2019-06-24 (Actual); Last update posted 2024-12-27 (Actual); Status verified 2024-12

CONDITIONS: Cerebral Arteriovenous Malformation
Keywords: arteriovenous malformation; MRI; DSA; Gamma Knife
MeSH Terms: conditions — Intracranial Arteriovenous Malformations; Arteriovenous Malformations

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
Cerebral arteriovenous malformations (AVMs) are abnormal vessels, connecting cerebral arteries and veins. They form a bundle which is called nidus. Rupture of an AVM leads to intracranial hemorrhage often causing neurological impairment or even death. As treatment can be associated with high rates of morbidity and mortality, AVMs still remain a considerable challenge for neurosurgeons. For smaller AVMs, a well-established treatment option is non-invasive Gamma Knife radiosurgery (GKRS). GKRS uses radiation to obliterate the AVM nidus hence, eliminating the risk of hemorrhage. However, after Gamma Knife radiosurgery, occlusion of the AVM nidus takes about two years. To evaluate treatment success after GKRS, invasive digital subtraction angiography (DSA) is still the gold standard. For this procedure, patients have to undergo puncture of the femoral artery for application of a contrast media to receive adequate imaging of the cerebral arteries. In recent literature it has been discussed whether sufficient evaluation of treatment is possible with non-invasive magnetic resonance imaging (MRI). At present, it is unclear whether this method could replace the current invasive gold standard for treatment evaluation. To investigate on this issue, a few studies have compared the two methods however, only retrospective data exist. Thus, the investigators are conducting this prospective study including 50 patients with cerebral AVMs treated with GRKS to evaluate the sensitivity for nidus obliteration of MRI using DSA as a reference.

DETAILED DESCRIPTION:
Background

Cerebral arteriovenous malformations consist of tangled blood vessels forming a so-called nidus which connects arteries to veins without the interposition of a capillary bed. Due to subsequent structural changes of draining veins within the nidus, patients are at risk of cerebral hemorrhage. Bleedings of AVMs are associated with high morbidity and mortality. Therefore, once a cerebral AVM is diagnosed, preventive treatment usually is aimed for. If hemorrhage already occurred treatment is necessary because of a high chance of re-bleeding. Cerebral AVMs are likely to cause neurological symptoms such as seizures and focal deficits without bleeding. These symptoms are usually due to the AVM's mass effect however, they have also been discussed to be caused by a vascular steal syndrome.

Etiology

The etiology of cerebral AVMs is not known. Aside from the possibility of a multifactorial cause it seems that genetic mutation and angiogenetic stimulation could play a role in their development. It is also discussed whether AVMs develop in utero or through an angiopathic reaction following ischemia or hemorrhage.

Epidemiology

The prevalence and incidence of cerebral AVMs are about 10 per 100,000 and 1 per 100,000; respectively without sex predilection. The annual risk of intracranial hemorrhage ranges from 1.2% in unruptured AVMs to 4.8% when hemorrhage already occurred before. The mortality rate among AVM patients after intracranial hemorrhage is 10-15%. The morbidity varies from 30-50%. Of all AVM patients without hemorrhage about 15-40% suffer from seizures. Progressive neurological deficit occurs at 6-12%.

Diagnosis

Cerebral AVMs are usually diagnosed by an MRI examination. They can easily be identified on enhanced images but may also be visible without contrast due to edema or mass effect. The current gold standard of diagnosis and evaluation of treatment success of cerebral AVMs is digital subtraction angiography (DSA). This method uses injection of a contrast agent into the patient's arteries and X-rays to visualize cerebral vessels. Imaging of the blood flow over time and therefore accurate distinction of feeding and draining vessels within the nidus is the major advantage of DSA. Subtraction of bones and soft tissue enables an optimal view of the vascular system.

DSA has to be carried out as an inpatient procedure because of its invasiveness. Occurrence of hematoma or pseudoaneurysm at the site of puncture and endovascular injury with consecutive embolism are rare but possible complications. Further disadvantages of DSA are a substantial exposure to radiation and the necessity of 24 hours of bed rest after the procedure which may lead to an increased risk of thrombosis.

Classification - The Spetzler-Martin grading-system

Evaluation of the Spetzler-Martin grade (SM grade) requires three characteristics of the AVM. first it is the size of the malformation regrouped into three categories. Next, the drainage is of importance: one can differentiate between superficial only and deep veins partaking in drainage. Finally, the eloquence of the brain tissue surrounding the lesion is considered. Areas responsible for higher functions such as movement and sensibility, vision and language are called eloquent. The thalamus, hypothalamus, brainstem and cerebellar peduncles are eloquent regions. On the cerebral cortex sensorimotor areas and those responsible for language and primary vision are eloquent.

The Spetzler-Martin system was developed to estimate the prognosis before surgical intervention, but is also used for other treatment methods. The SM grade correlates well with the difficulty of surgery and its outcome.

Treatment

There are different treatment options for cerebral AVMs: Microsurgical resection, endovascular embolization and Gamma Knife radiosurgery, or combinations thereof. Independent of AVM specifications and treatment option, any therapy bears the risk of cerebral hemorrhage and ischemia and therefore permanent neurological deficit and death. Hence, the decision if and how an AVM should be treated has to be made carefully with the intention to offer a result better than the natural course of the disease. In order to answer the question if a wait-and-see strategy is a valid option, a prospective, non-blinded, randomized, multicenter study was conducted in 2014. The study compared the risk of death and stroke as well as functional outcome between treated and untreated AVM patients.

The so-called ARUBA trial was interrupted six years after the beginning of randomization due to an apparent superiority of the untreated group. The authors concluded that unruptured cerebral AVMs should be managed conservatively.The study was harshly criticized by many experts due to its setting and the interpretation of the data. One major limitation is that different treatment options were not evaluated separately but as one interventional group. Other limitations of ARUBA are a low number of cases - only 116 patients were randomized for intervention and of those only five underwent microsurgical resection - and a short follow-up of 33 months. At least, ARUBA shows the controversy existing among experts concerning cerebral AVM treatment. The established treatment options will be explained below.

Microsurgical Resection

As microsurgical resection eliminates the risk of bleeding immediately, it still represents the therapy of choice for most of the cerebral AVMs reaching a Spetzler-Martin score of one to three. In order to expose a cerebral AVM, a bone flap of the patient's skull is raised and the dura opened. Feeders are identified, coagulated and cut so the AVM can be resected in total. Outcome of patients with an unruptured AVM undergoing microsurgery depends on their Spetzler-Martin (SM) grade. According to a prospective cohort study from 2014 a permanent neurological deficit is postoperatively seen in 1.6% of patients with SM scores 1 and 2. In patient with SM grade 3 the risk of permanent neurological deficit after surgery rises to 14.0% and to 38.6% in patients with SM grades 4 and 5.

Endovascular Embolization

Endovascular embolization of an AVM is performed via the arterial route after puncture of a peripheral artery. The AVM nidus is occluded by injection of an embolic material which clogs its feeding arteries. According to a systematic review including more than 1,000 AVM patients who had undergone endovascular embolization, this therapy lead to nidus occlusion in an average of 13%, with a wide range from 0 to 94%. Permanent neurological deficit after embolization was averagely seen in 6.6%, ranging from 0 to 28%. The endovascular approach is often used to close small AVMs or to make larger AVMs amenable for radiosurgery or microsurgery.

Gamma Knife Radiosurgery

Gamma Knife Radiosurgery can be performed either as a single therapy or in combination with other treatment methods, most commonly combined with endovascular embolization. At the Department of Neurosurgery, MUV radiosurgery of cerebral AVMs is performed with Gamma Knife Perfexion® which uses 192 cobalt 60 sources to apply high dose radiation into an exactly defined volume within the cranium. Gamma Knife radiosurgery is generally performed in local anesthesia thus enabling the fixation of the stereotactic frame to the skull. In children below 14 years of age Gamma Knife radiosurgery is performed under general anesthesia. Whereas endovascular and surgical treatment immediately eliminate the risk of bleeding if carried out successfully, nidus occlusion after Gamma Knife radiosurgery usually takes about two years. During this time the bleeding risk is reported to be the same as in untreated patients. The major advantage of radiosurgery is its non-invasiveness. Rates of complete nidus occlusion after Gamma Knife radiosurgery of cerebral AVMs are reported to be about 85% for AVMs with a SM grade 1 to 3. A much lower rate of 54% for AVMs with a SM grade 4 and a rate of 0% for AVMs with SM grade 5 show the dependence of the Spetzler-Martin grade. However, even if nidus occlusion is not achieved in many AVMs with higher SM grade, a reduction of their size may enable further treatment. Permanent neurological deficit after radiosurgery was seen in 5.1% with a range from 0 to 21%.23 Complications of radiosurgery are adverse radiation effects (ARE) which occur many years after intervention and include perilesional edema and cyst formation. Those have to be differentiated from radiation induced changes (RIC) arising in the first 1-2 years after treatment and including focal necrosis, white matter injury, microangiopathy, sinus inflammation and atrophy.

Treatment Evaluation

The gold standard for the evaluation after AVM therapy is the catheter angiography; digital subtraction angiography (DSA). As already mentioned in chapter Diagnosis, DSA has several disadvantages like invasiveness, necessity of inpatient treatment and peri-interventional risks. So far, MRI/MRA is a regularly performed evaluation method after Gamma Knife treatment of AVMs but it still remains unclear if its accuracy is sufficient compared to that of DSA. Numerous MRI protocols for imaging of cerebral vascular pathologies exist. According to a small prospective study a specific MRI protocol focusing on blood flow characteristics called arterial spin labeling (ASL) was superior to conventional contrast enhanced MRI in the evaluation of AVM nidus occlusion after stereotactic radiosurgery. Using DSA as a reference, seven out of seven patients with complete nidus occlusion where assessed correctly by ASL imaging, so were three patients with a persisting AVM nidus.

However, in those three cases, according to the contrast enhanced MRI the nidus was falsely rated as occluded. A retrospective study comparing conventional MRI/MRA to DSA found 80% sensitivity and 90% specificity of standard MRI/MRA for detection of AVM nidus occlusion after stereotactic radiosurgery in a series of 136 patients.

Objectives and hypotheses

Objective:

To evaluate sensitivity and specificity of a standardized MRI/MRA protocol compared to that of DSA for detection of nidus occlusion after Gamma Knife radiosurgery of cerebral AVMs

Hypotheses:

H0: There is significant difference in sensitivity and specificity between MRI/MRA and DSA for detection of nidus occlusion after Gamma Knife radiosurgery of cerebral AVMs.

H1: There is no significant difference in sensitivity and specificity between MRI/MRA and DSA for detection of nidus occlusion after Gamma Knife radiosurgery of cerebral AVMs.

Methods

In this preliminary study the investigators plan to include about 50 radiosurgically treated patients with cerebral AVMs. Patients participating in the study will not be exposed to any additional risk compared to patients not participating in the study. Participants will undergo a standardized MRI protocol at the Department of Radiology, MUV two years after Gamma Knife treatment. The standardized MRI protocol replaces the follow-up-MRI two years after treatment that is usually performed in private practice and often does not include all required sequences. The standardized MRI protocol includes specific sequences allowing analyzation of vascular pathologies. Those are a contrast enhanced three-dimensional MRA (T1 GE 3D +/- KM), a time-of-flight magnetic resonance angiography (TOF-MRA), arterial spin labeling (ASL) and time resolved MRA with interleaved stochastic trajectories (TWIST-MRA). Three dimensional MRA and TOF-MRA produce conventional images of vascular structures. ASL enables more detailed imaging of the cerebral blood flow. TWIST-MRA produces time resolved images. Hence, the major advantage of DSA should be reproduced with this method.

For evaluation of the parenchyma adjacent to the AVM, DWI and SWI sequences will allow detection of ischemic areas and hemorrhage. Standard sequences (T2 sagittal, axial and coronal) will also be produced. Participants of this study will be enrolled at the Gamma Knife outpatient clinic of the Department of Neurosurgery, MUV. Nidus occlusion will be evaluated by a neuroradiologist and compared to the gold standard of DSA performed at the Department of Neurosurgery, MUV. Since the angiography (DSA) is the current gold standard in AVM evaluation it will be performed in any case and is thus rated as outside of this study protocol. Thus, sensitivity and specificity of MRI/MRA for detection of AVM nidus occlusion will be assessed in comparison to the gold standard. Due to the fact that every case of cerebral AVM treated by stereotactic radiosurgery at the Department of Neurosurgery, Medical University of Vienna is assessed by MRI and DSA examinations after treatment, the post-radiosurgical procedures of diagnosis do not pose any additional effort or risk for patients participating in the study. In fact, patients may benefit from participation as they do not need to care for scheduling of their MRI examination in private practice.

Statistical analysis

Due to an uneven distribution of data, statistical analysis will be performed with nonparametric tests. Descriptive analysis of characteristics of patients and AVMs as well as Gamma Knife parameters includes the median value and range as well as frequencies, numbers and percentages. Statistical calculations for comparison between eventual treatment groups include the Kruskal-Wallis, Mann-Whitney-U and Chi-square test for independent samples. To support the hypothesis, the result of the MRI examination must be in accordance with the result of the DSA examination in a vast majority of cases. The investigators set a 95% threshold for the sensitivity of MRI examinations to be sufficient for confirming the hypothesis in this preliminary setting. Relevant findings have to be confirmed in a larger (multicenter) prospective study.

Sample size

The approximate sample size of 50 patients is due to the planned study duration of 3 years. The study serves as a preliminary study and results may be confirmed by a larger (multicenter) study.

Recruiting of patients

Patients will be recruited in the Gamma Knife outpatient clinic of the Department of Neurosurgery, MUV. Patients must undergo or have undergone Gamma Knife radiosurgery due to cerebral AVM. For inclusion patients must have their two-year follow-up MRI exam within the duration of study. All patients have to sign a form for participation in the study after purpose and process of the study has been explained to them. The investigators plan to enroll about 50 patients for this study.

Quality and protection of data

Entry and handling of patient data will only be executed by trained medical staff involved in the planning and conduction of the study. Patient data will be entered anonymized in a SPSS file using IBM SPSS Statistics for Windows (Version 25.0 Armonk, NY: IBM Corp.).

Variables used in the registry

Patient sex: male/female Source: EDP system

Patient age: years Source: EDP system

AVM diameter: cm Source: pre-radiosurgical MRI

AVM localization: frontal, parietal, occipital, temporal, insular, limbic, cerebellar, brain stem, basal ganglia, thalamus, intraventricular, corpus callosum Source: pre-radiosurgical MRI

Number of AVM feeders: Number Source: pre-radiosurgical DSA

AVM-haemorrhage: Yes/No Source: Anamnesis in EDP system

RBAS (Modified Radiosurgery Based AVM score): <1 to >2 Source: Pre-radiosurgical MRI

VRAS (Virginia Radiosurgery AVM Scale): 0 to 4 points

Treatment: Radiosurgery only, Radiosurgery+Endovascular embolization, other combinations including Radiosurgery Source: EDP system

Date of treatment: Date Source: EDP system

Gamma Knife parameters: Isodose (%), Marginal dose (Gy), Maximum dose (Gy), Radiation volume (ccm) Source: EDP system

Substance for embolization in case of additional endovascular treatment to radiosurgery: Histoacryl, Onyx, ethanol, coils, cyanoacrylate, Glubran

ELIGIBILITY:
Inclusion Criteria:

* Patients must undergo or have undergone Gamma Knife radiosurgery due to cerebral AVM
* For inclusion patients must have their two-year follow-up MRI exam within the duration of study
* All patients have to sign a form for participation in the study after purpose and process of the study has been explained to them.
* For patients younger than 18 years, a parent or legal guardian has to sign a form for participation after being informed about purpose and process of the study have been explained to them.

Exclusion Criteria:

* Patients who do not give informed consent to participate
* Patients younger than 16 years

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients must undergo or have undergone Gamma Knife radiosurgery due to cerebral AVM at the Department of Neurosurgery, Medical University of Vienna. For inclusion patients must have their two-year follow-up MRI exam within the duration of study.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-07-01 (Actual); Primary Completion 2024-07-01 (Actual); Study Completion 2024-10-01 (Actual)

PRIMARY OUTCOMES:
Post radiosurgical AVM nidus obliteration on MRI | The MRI examination will be performed 2 years after Gamma Knife treatment.
  Sensitivity and specificity of MRI/MRA evaluated by catheter angiography
Post radiosurgical AVM nidus obliteration on DSA | DSA will be performed within 2 months after MRI/MRA
  Reference method for evaluation of sensitivity and specificity of MRI/MRA

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Neurosurgery, Medical University of Vienna, Vienna, Austria

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fleetwood IG, Steinberg GK. Arteriovenous malformations. Lancet. 2002 Mar 9;359(9309):863-73. doi: 10.1016/S0140-6736(02)07946-1. PMID 11897302
- [Background] Gross BA, Du R. Natural history of cerebral arteriovenous malformations: a meta-analysis. J Neurosurg. 2013 Feb;118(2):437-43. doi: 10.3171/2012.10.JNS121280. Epub 2012 Nov 30. PMID 23198804
- [Background] Friedlander RM. Clinical practice. Arteriovenous malformations of the brain. N Engl J Med. 2007 Jun 28;356(26):2704-12. doi: 10.1056/NEJMcp067192. No abstract available. PMID 17596605
- [Background] Mullan S, Mojtahedi S, Johnson DL, Macdonald RL. Embryological basis of some aspects of cerebral vascular fistulas and malformations. J Neurosurg. 1996 Jul;85(1):1-8. doi: 10.3171/jns.1996.85.1.0001. PMID 8683257
- [Background] Lasjaunias P. A revised concept of the congenital nature of cerebral arteriovenous malformations. Interv Neuroradiol. 1997 Dec 20;3(4):275-81. doi: 10.1177/159101999700300401. Epub 2001 May 15. PMID 20678357
- [Background] Berman MF, Sciacca RR, Pile-Spellman J, Stapf C, Connolly ES Jr, Mohr JP, Young WL. The epidemiology of brain arteriovenous malformations. Neurosurgery. 2000 Aug;47(2):389-96; discussion 397. doi: 10.1097/00006123-200008000-00023. PMID 10942012
- [Background] Derdeyn CP, Zipfel GJ, Albuquerque FC, Cooke DL, Feldmann E, Sheehan JP, Torner JC; American Heart Association Stroke Council. Management of Brain Arteriovenous Malformations: A Scientific Statement for Healthcare Professionals From the American Heart Association/American Stroke Association. Stroke. 2017 Aug;48(8):e200-e224. doi: 10.1161/STR.0000000000000134. Epub 2017 Jun 22. PMID 28642352
- [Background] Graf CJ, Perret GE, Torner JC. Bleeding from cerebral arteriovenous malformations as part of their natural history. J Neurosurg. 1983 Mar;58(3):331-7. doi: 10.3171/jns.1983.58.3.0331. PMID 6827317
- [Background] Leblanc R, Levesque M, Comair Y, Ethier R. Magnetic resonance imaging of cerebral arteriovenous malformations. Neurosurgery. 1987 Jul;21(1):15-20. doi: 10.1227/00006123-198707000-00004. PMID 3614598
- [Background] Shankar JJ, Lum C, Chakraborty S, Dos Santos M. Cerebral vascular malformations: Time-resolved CT angiography compared to DSA. Neuroradiol J. 2015 Jun;28(3):310-5. doi: 10.1177/1971400915589682. PMID 26246101
- [Background] Yoon W, Kim H, Kim YW, Kim SR, Park IS. Usefulness and Stability of Intraoperative Digital Subtraction Angiography Using the Transradial Route in Arteriovenous Malformation Surgery. World Neurosurg. 2018 Mar;111:e799-e805. doi: 10.1016/j.wneu.2017.12.164. Epub 2018 Jan 5. PMID 29309977
- [Background] Spetzler RF, Martin NA. A proposed grading system for arteriovenous malformations. J Neurosurg. 1986 Oct;65(4):476-83. doi: 10.3171/jns.1986.65.4.0476. PMID 3760956
- [Background] Hamilton MG, Spetzler RF. The prospective application of a grading system for arteriovenous malformations. Neurosurgery. 1994 Jan;34(1):2-6; discussion 6-7. PMID 8121564
- [Background] Morgan MK, Sekhon LH, Finfer S, Grinnell V. Delayed neurological deterioration following resection of arteriovenous malformations of the brain. J Neurosurg. 1999 Apr;90(4):695-701. doi: 10.3171/jns.1999.90.4.0695. PMID 10193615
- [Background] Lunsford LD, Niranjan A, Kano H, Kondziolka D. The technical evolution of gamma knife radiosurgery for arteriovenous malformations. Prog Neurol Surg. 2013;27:22-34. doi: 10.1159/000341625. Epub 2012 Dec 11. PMID 23258506
- [Background] van Beijnum J, van der Worp HB, Buis DR, Al-Shahi Salman R, Kappelle LJ, Rinkel GJ, van der Sprenkel JW, Vandertop WP, Algra A, Klijn CJ. Treatment of brain arteriovenous malformations: a systematic review and meta-analysis. JAMA. 2011 Nov 9;306(18):2011-9. doi: 10.1001/jama.2011.1632. PMID 22068993
- [Background] Peschillo S, Delfini R. Endovascular neurosurgery in Europe and in Italy: what is in the future? World Neurosurg. 2012 Feb;77(2):248-51. doi: 10.1016/j.wneu.2011.05.055. Epub 2011 Nov 7. PMID 22120373
- [Background] Ogilvy CS, Stieg PE, Awad I, Brown RD Jr, Kondziolka D, Rosenwasser R, Young WL, Hademenos G; Special Writing Group of the Stroke Council, American Stroke Association. AHA Scientific Statement: Recommendations for the management of intracranial arteriovenous malformations: a statement for healthcare professionals from a special writing group of the Stroke Council, American Stroke Association. Stroke. 2001 Jun;32(6):1458-71. doi: 10.1161/01.str.32.6.1458. No abstract available. PMID 11387517
- [Background] Mohr JP, Parides MK, Stapf C, Moquete E, Moy CS, Overbey JR, Al-Shahi Salman R, Vicaut E, Young WL, Houdart E, Cordonnier C, Stefani MA, Hartmann A, von Kummer R, Biondi A, Berkefeld J, Klijn CJ, Harkness K, Libman R, Barreau X, Moskowitz AJ; international ARUBA investigators. Medical management with or without interventional therapy for unruptured brain arteriovenous malformations (ARUBA): a multicentre, non-blinded, randomised trial. Lancet. 2014 Feb 15;383(9917):614-21. doi: 10.1016/S0140-6736(13)62302-8. Epub 2013 Nov 20. PMID 24268105
- [Background] Meling TR, Proust F, Gruber A, Niemela M, Regli L, Roche PH, Vajkoczy P. On apples, oranges, and ARUBA. Acta Neurochir (Wien). 2014 Sep;156(9):1775-9. doi: 10.1007/s00701-014-2140-7. Epub 2014 Jun 3. No abstract available. PMID 24890935
- [Background] Bervini D, Morgan MK, Ritson EA, Heller G. Surgery for unruptured arteriovenous malformations of the brain is better than conservative management for selected cases: a prospective cohort study. J Neurosurg. 2014 Oct;121(4):878-90. doi: 10.3171/2014.7.JNS132691. Epub 2014 Aug 8. PMID 25105704
- [Background] Plasencia AR, Santillan A. Embolization and radiosurgery for arteriovenous malformations. Surg Neurol Int. 2012;3(Suppl 2):S90-S104. doi: 10.4103/2152-7806.95420. Epub 2012 Apr 26. PMID 22826821
- [Background] Kano H, Kondziolka D, Flickinger JC, Yang HC, Flannery TJ, Awan NR, Niranjan A, Novotny J Jr, Lunsford LD. Stereotactic radiosurgery for arteriovenous malformations, Part 3: outcome predictors and risks after repeat radiosurgery. J Neurosurg. 2012 Jan;116(1):21-32. doi: 10.3171/2011.9.JNS101741. Epub 2011 Nov 11. PMID 22077445
- [Background] Koltz MT, Polifka AJ, Saltos A, Slawson RG, Kwok Y, Aldrich EF, Simard JM. Long-term outcome of Gamma Knife stereotactic radiosurgery for arteriovenous malformations graded by the Spetzler-Martin classification. J Neurosurg. 2013 Jan;118(1):74-83. doi: 10.3171/2012.9.JNS112329. Epub 2012 Oct 19. PMID 23082882
- [Background] Kano H, Flickinger JC, Tonetti D, Hsu A, Yang HC, Flannery TJ, Niranjan A, Lunsford LD. Estimating the Risks of Adverse Radiation Effects After Gamma Knife Radiosurgery for Arteriovenous Malformations. Stroke. 2017 Jan;48(1):84-90. doi: 10.1161/STROKEAHA.116.014825. Epub 2016 Nov 29. PMID 27899758
- [Background] Lee CC, Reardon MA, Ball BZ, Chen CJ, Yen CP, Xu Z, Wintermark M, Sheehan J. The predictive value of magnetic resonance imaging in evaluating intracranial arteriovenous malformation obliteration after stereotactic radiosurgery. J Neurosurg. 2015 Jul;123(1):136-44. doi: 10.3171/2014.10.JNS141565. Epub 2015 Apr 3. PMID 25839923
- [Background] Deutschmann HA, Augustin M, Simbrunner J, Unger B, Schoellnast H, Fritz GA, Klein GE. Diagnostic accuracy of 3D time-of-flight MR angiography compared with digital subtraction angiography for follow-up of coiled intracranial aneurysms: influence of aneurysm size. AJNR Am J Neuroradiol. 2007 Apr;28(4):628-34. PMID 17416811
- [Background] Huang X, Zhou S, Su T, Ye L, Zhu PW, Shi WQ, Min YL, Yuan Q, Yang QC, Zhou FQ, Shao Y. Resting cerebral blood flow alterations specific to the comitant exophoria patients revealed by arterial spin labeling perfusion magnetic resonance imaging. Microvasc Res. 2018 Nov;120:67-73. doi: 10.1016/j.mvr.2018.06.007. Epub 2018 Jul 2. PMID 29991447
- [Background] Hammer S, Uller W, Manger F, Fellner C, Zeman F, Wohlgemuth WA. Time-resolved magnetic resonance angiography (MRA) at 3.0 Tesla for evaluation of hemodynamic characteristics of vascular malformations: description of distinct subgroups. Eur Radiol. 2017 Jan;27(1):296-305. doi: 10.1007/s00330-016-4270-1. Epub 2016 Feb 23. PMID 26905867
- [Background] Kodera T, Arai Y, Arishima H, Higashino Y, Isozaki M, Tsunetoshi K, Matsuda K, Kitai R, Shimizu K, Kosaka N, Yamamoto T, Shioura H, Kimura H, Kikuta KI. Evaluation of obliteration of arteriovenous malformations after stereotactic radiosurgery with arterial spin labeling MR imaging. Br J Neurosurg. 2017 Dec;31(6):641-647. doi: 10.1080/02688697.2017.1365818. Epub 2017 Aug 22. PMID 28830253
- [Background] Higgins LJ, Koshy J, Mitchell SE, Weiss CR, Carson KA, Huisman TA, Tekes A. Time-resolved contrast-enhanced MRA (TWIST) with gadofosveset trisodium in the classification of soft-tissue vascular anomalies in the head and neck in children following updated 2014 ISSVA classification: first report on systematic evaluation of MRI and TWIST in a cohort of 47 children. Clin Radiol. 2016 Jan;71(1):32-9. doi: 10.1016/j.crad.2015.09.006. Epub 2015 Oct 21. PMID 26474946